CLINICAL TRIAL: NCT01885936
Title: A Phase 1/2 Double-Blind Study of the Safety and Efficacy of Albuterol on Motor Function in Individuals With Late-onset Pompe Disease Receiving Enzyme Replacement Therapy
Brief Title: Safety and Efficacy of Albuterol in Individuals With Late-onset Pompe Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00046020
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pompe Disease
Keywords: LOPD; Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol (Experimental): Initially 4 mg daily for one week, then 4 mg BID per oral daily for the next 5 weeks. If the 4 mg BID per oral is well tolerated, the dose will be increased to 8 mg each morning/4 mg each evening for one week, followed by 8 mg BID per oral for the remainder of the study.
  Interventions: Drug: Albuterol
- Placebo Comparator (Placebo Comparator): Initially one capsule daily for one week, then one capsule BID per oral daily for the next 5 weeks. If the one capsule BID per oral is well tolerated, the dose will be increased to two capsules each morning/one capsule each evening for one week, followed by two capsules BID per oral for the remainder of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albuterol — Initially 4 mg daily for one week, 4 mg BID per oral daily for the next 5 weeks. If the 4 mg BID per oral is well tolerated, the dose will be increased to 8 mg each morning/4 mg each evening for one week, followed by 8 mg BID per oral for the remainder of the study.
  Arms: Albuterol
Drug: Placebo — Initially one capsule daily for one week, then one capsule BID per oral daily for the next 5 weeks. If the one capsule BID per oral is well tolerated, the dose will be increased to two capsules each morning/one capsule each evening for one week, followed by two capsules BID per oral for the remainder of the study.
  Arms: Placebo Comparator

SUMMARY:
In this study the study team proposes to investigate the efficacy of albuterol on motor function of individuals with Late Onset Pompe Disease (LOPD) who are receiving enzyme replacement therapy, given albuterol was well-tolerated in patients with Late Onset Pompe Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Pompe disease by blood acid alpha-glucosidase assay and acid alpha-glucosidase gene sequencing,
2. Age: 18+ years at enrollment.
3. Receiving enzyme replacement therapy at standard dose (20 mg/kg every 2 weeks) for at least 52 weeks.
4. Subjects are capable of giving written consent.

Exclusion Criteria:

1. Continuous invasive ventilation (via tracheostomy or endotracheal tube).
2. Clinically relevant illness within two weeks of enrollment including fever > 38.2 C, vomiting more than once in 24 hours, seizure, or other symptom deemed contraindicative to new therapy.
3. Chronic heart disease (Myocardial infarction in the past 2 months, arrhythmia, cardiomyopathy).
4. History of seizure disorder.
5. History of diabetes.
6. Hypokalemia.
7. History of hyperthyroidism.
8. Pregnancy.
9. Patients on a non-standard schedule for enzyme replacement therapy; for example, weekly infusions as opposed to infusions every two weeks.
10. Anti-rhGAA antibody titer > 1:100,000
11. History of hypersensitivity to Beta 2-agonist drugs such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline, salmeterol (Serevent)..
12. The use of the following medications:

    * diuretics (water pill);
    * digoxin (digitalis, Lanoxin);
    * beta-blockers such as atenolol (Tenormin), metoprolol (Lopressor), and propranolol (Inderal);
    * tricyclic antidepressants such as amitriptyline (Elavil, Etrafon), doxepin (Sinequan), imipramine (Janimine, Tofranil), and nortriptyline (Pamelor);
    * Monoamine oxidase inhibitors such as isocarboxazid (Marplan), phenelzine (Nardil), rasagiline (Azilect), selegiline (Eldepryl, Emsam), or tranylcypromine (Parnate); or
    * bronchodilators such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline (Brethine, Bricanyl), salmeterol (Serevent), isoetharine (Bronkometer), metaproterenol (Alupent, Metaprel), or isoproterenol (Isuprel Mistometer) within 12 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dwight d Koeberl, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koeberl DD, Li S, Dai J, Thurberg BL, Bali D, Kishnani PS. beta2 Agonists enhance the efficacy of simultaneous enzyme replacement therapy in murine Pompe disease. Mol Genet Metab. 2012 Feb;105(2):221-7. doi: 10.1016/j.ymgme.2011.11.005. Epub 2011 Nov 11. PMID 22154081
- [Derived] Koeberl DD, Case LE, Desai A, Smith EC, Walters C, Han SO, Thurberg BL, Young SP, Bali D, Kishnani PS. Improved muscle function in a phase I/II clinical trial of albuterol in Pompe disease. Mol Genet Metab. 2020 Feb;129(2):67-72. doi: 10.1016/j.ymgme.2019.12.008. Epub 2019 Dec 10. PMID 31839530

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three enrolled participants decided to withdraw due to travel difficulties.
Groups:
- Albuterol: Initially 4 mg daily for one week, 4 mg BID (twice a day) per oral for the next 5 weeks. If the 4 mg BID per oral is well tolerated, the dose will be increased to 8 mg each morning/4 mg each evening for one week, followed by 8 mg BID per oral for the remainder of the study.
- Placebo Comparator: Placebo administered
Period: Overall Study
Arm/Group | Albuterol | Placebo Comparator
Started | 8 | 5
Completed | 7 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol | Placebo Comparator | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (9.7) | 53.4 (9.9) | 49.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Description: All participants who experienced adverse events.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Albuterol | Placebo Comparator
Number analyzed (Participants) | 8 | 5
Participants | 5 | 5

2. Secondary Outcome: Change in Forced Vital Capacity From Pulmonary Function Tests at 30 Weeks and 52 Weeks.
Description: FVC (forced vital capacity) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Week 30, and Week 52
Population: One subject dropped out from the albuterol group. Later participants were unblinded and switched to drug before Week 52 under an IRB (Institutional Review Board) approved amendment, and 4 late-enrolled drug and 3 late-enrolled placebo subjects could not be included in the analysis at Week 52.
Measure: Mean (Standard Deviation); unit: Percent of predicted FVC
Arm/Group | Albuterol | Placebo Comparator
Number analyzed (Participants) | 7 | 5
Percent of predicted FVC
  Change at 30 Weeks | -0.2 (5.7) | 0.4 (7.9)
  Change at 52 Weeks: number analyzed (Participants) | 3 | 2
  Change at 52 Weeks | -1.3 (6.2) | 3.0 (5.7)

3. Secondary Outcome: Change in 6 Minute Walk Test
Description: The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. Assessed by physical therapist.
Time Frame: Baseline, Week 6, and Week 52
Population: Early participants were not randomized until 6 weeks; 3 drug and 2 placebo subjects could not be included in the analysis. One drug subject missed the Week 6 visit, and one placebo subject could not perform the 6 minute walk test. Later participants were unblinded before Week 52. Four drug and 3 placebo subjects could not be included at Week 52.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Albuterol | Placebo Comparator
Number analyzed (Participants) | 3 | 2
meters
  Change at 6 Weeks | 24.0 (10.3) | 32.0 (58.1)
  Change at 52 Weeks | 43.6 (26.0) | 13.6 (0.9)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Arm/Group | Albuterol | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 5/8 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol (N=8) | Placebo Comparator (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ankle edema increase (Cardiac disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Body aches (Musculoskeletal and connective tissue disorders) | 0 | 2
Body cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain fog (Nervous system disorders) | 1 | 0
Chest tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dry eyes (Eye disorders) | 1 | 0
Dry mucous membranes (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Energy decrease (General disorders) | 0 | 1
Fall (General disorders) | 1 | 4
Fatigue (General disorders) | 2 | 0
Fever (General disorders) | 1 | 0
Foot cramps (Musculoskeletal and connective tissue disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Hand cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 1
Hypertension (Cardiac disorders) | 0 | 1
Insomnia (General disorders) | 5 | 1
Jaw cramps (Musculoskeletal and connective tissue disorders) | 2 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 4 | 1
Otitis (Ear and labyrinth disorders) | 2 | 0
Pain (Nervous system disorders) | 3 | 5
Palpitations (Cardiac disorders) | 3 | 2
Peripheral neuropathy increase (Nervous system disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shortness of breath (General disorders) | 1 | 0
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (General disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 4 | 0
Throat cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1
Tremors (General disorders) | 2 | 0
Urination increase (Renal and urinary disorders) | 3 | 0
Weight gain (General disorders) | 1 | 0
Weight loss (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes